CLINICAL TRIAL: NCT02684955
Title: Non-invasive Neurological Evaluation During Cardiopulmonary Resuscitation for Out of Hospital Cardiac Arrest Patients Neuro-E-CPR Study
Brief Title: Non-invasive Neurological Evaluation During CPR
Acronym: Neuro-E-CPR
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: Neuro-E-CPR
Record Dates: First submitted 2016-02-09; First posted 2016-02-18 (Estimated); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Cardiac Arrest
Keywords: cardiac arrest; near-infrared spectroscopy; automated infrared pupillometry; prognostication
MeSH Terms: conditions — Heart Arrest | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cerebral spectroscopy + pupillometry: During CPR, rSO2 will be monitored continuously as well as quantitative measurements of the pupillary light reaction every 5 minutes.
  Interventions: Device: Cerebral spectroscopy; Device: Pupillometry

INTERVENTIONS:
Device: Cerebral spectroscopy — Cerebral spectroscopy (near-infrared spectroscopy - NIRS) allows to measure with a noninvasive method the local oxygen saturation of the prefrontal cortex (rSO2), reflecting the balance between need and supply of brain oxygenation.
  Other Names: near-infrared spectroscopy - NIRS
Device: Pupillometry — The quantitative measurement of the pupillary light reaction has been described to predict neurological outcome

SUMMARY:
Cardiac arrest remains a leading cause of death, currently affecting >250,000 Europeans outside the hospital each year. Manual cardiopulmonary resuscitation (CPR) provides between 15 to 30 % of normal blood flow to the heart and brain. For out-of-hospital cardiac arrest, the return of spontaneous circulation (ROSC) is possible only for 20-40% of patients with trained resuscitation teams. However, only 5-10% of patients will survive with good neurological status. A good quality CPR, a short time before initiation of the resuscitation and a short delay before the first defibrillation have been associated with improved neurological outcome. Unfortunately it is currently impossible to obtain reliable information on the quality of the perfusion and oxygenation of organs during CPR. The current monitoring during CPR is limited to heart rhythm analysis, pulse rate evaluation and end tidal CO2 (EtCO2). The last one is the only parameter which have been linked with probability of ROSC and its value gives no indication of the long-term prognosis nor the neurological status.

Cerebral spectroscopy (near-infrared spectroscopy - NIRS) allows to measure with a noninvasive method the local oxygen saturation of the prefrontal cortex (rSO2), reflecting the balance between need and supply of brain oxygenation. This technique has been recently used in cardiac arrest showing a possible association between rSO2 measured during CPR and the occurrence of ROSC or survival. The quantitative measurement of the pupillary light reaction has been described to predict neurological outcome in the hospital for patient successfully reanimated after out-of-hospital cardiac arrest (OHCA). Recently, a feasibility study has shown that its use was also possible during CPR in the pre-hospital setting.

The investigators aim to study a composite prognostic factor combining quantitative rSO2 and automated pupillometry measured during CPR. The investigators hypothesized that the rate of survival with good neurologic outcome at 30 days will be lower in patients with rSO2 <30% for more than 5 min and an absent pupillary reflex more than 5 min or decreasing during CPR .

ELIGIBILITY:
Inclusion Criteria:

* All adults with nontraumatic, out-of-hospital cardiac arrest

Exclusion Criteria:

* Traumatic cardiac arrest
* Patients who had achieved ROSC before inclusion patients with a do-not-attempt resuscitation order
* Patients < 18 years old
* Subjects known to be pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Out of Hospital cardiac arrest patient
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2016-02-09 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2019-08-22 (Actual)

PRIMARY OUTCOMES:
Prognostic value of rSO2, pupillometry, bystander CPR and initial cardiac rhythm alone or in association for survival at hospital admission | Through out-of-hospital care, an average of 2 hours
  rSO2, pupillometry, bystander CPR

SECONDARY OUTCOMES:
prognostic value of capnography alone or in association with primary outcomes parameters for survival at hospital admission | Through out-of-hospital care, an average of 2 hours
  EtCO2

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Savary, MD, Principal Investigator — Annecy Hospital
Locations (2):
- France (2):
  - SAMU 74, Annecy
  - SAMU 38, Grenoble

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Levine RL, Wayne MA, Miller CC. End-tidal carbon dioxide and outcome of out-of-hospital cardiac arrest. N Engl J Med. 1997 Jul 31;337(5):301-6. doi: 10.1056/NEJM199707313370503. PMID 9233867
- [Background] Storm C, Leithner C, Krannich A, Wutzler A, Ploner CJ, Trenkmann L, von Rheinbarben S, Schroeder T, Luckenbach F, Nee J. Regional cerebral oxygen saturation after cardiac arrest in 60 patients--a prospective outcome study. Resuscitation. 2014 Aug;85(8):1037-41. doi: 10.1016/j.resuscitation.2014.04.021. Epub 2014 Apr 30. PMID 24795284
- [Background] Ito N, Nishiyama K, Callaway CW, Orita T, Hayashida K, Arimoto H, Abe M, Endo T, Murai A, Ishikura K, Yamada N, Mizobuchi M, Anan H, Okuchi K, Yasuda H, Mochizuki T, Tsujimura Y, Nakayama T, Hatanaka T, Nagao K; J-POP Registry Investigators. Noninvasive regional cerebral oxygen saturation for neurological prognostication of patients with out-of-hospital cardiac arrest: a prospective multicenter observational study. Resuscitation. 2014 Jun;85(6):778-84. doi: 10.1016/j.resuscitation.2014.02.012. Epub 2014 Mar 5. PMID 24606889
- [Background] Singer AJ, Ahn A, Inigo-Santiago LA, Thode HC Jr, Henry MC, Parnia S. Cerebral oximetry levels during CPR are associated with return of spontaneous circulation following cardiac arrest: an observational study. Emerg Med J. 2015 May;32(5):353-6. doi: 10.1136/emermed-2013-203467. Epub 2014 Mar 24. PMID 24662518
- [Background] Schewe JC, Thudium MO, Kappler J, Steinhagen F, Eichhorn L, Erdfelder F, Heister U, Ellerkmann R. Monitoring of cerebral oxygen saturation during resuscitation in out-of-hospital cardiac arrest: a feasibility study in a physician staffed emergency medical system. Scand J Trauma Resusc Emerg Med. 2014 Oct 5;22:58. doi: 10.1186/s13049-014-0058-y. PMID 25286829
- [Background] Suys T, Bouzat P, Marques-Vidal P, Sala N, Payen JF, Rossetti AO, Oddo M. Automated quantitative pupillometry for the prognostication of coma after cardiac arrest. Neurocrit Care. 2014 Oct;21(2):300-8. doi: 10.1007/s12028-014-9981-z. PMID 24760270
- [Background] Behrends M, Niemann CU, Larson MD. Infrared pupillometry to detect the light reflex during cardiopulmonary resuscitation: a case series. Resuscitation. 2012 Oct;83(10):1223-8. doi: 10.1016/j.resuscitation.2012.05.013. Epub 2012 May 30. PMID 22659054